CLINICAL TRIAL: NCT03408925
Title: Preventing Lower Extremity Injury in Elite Orienteerers
Brief Title: Preventing Injury in Elite Orienteerers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Philip von Rosen, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-1645/2017
Record Dates: First submitted 2018-01-16; First posted 2018-01-24 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Lower Extremity Injury
Keywords: elite orienteering
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: RCT, two groups (intervention/control)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Test assessors and data collectors will be blinded to treatment allocation. The randomized phase will be unblinded after 14 weeks of data collection and the long-term follow-up (4 months) will be conducted by test assessors blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention consists of an exercise program developed by the medical team of the National Federation of Orienteering. Specifically, it consists of four exercises targeting strength, flexibility and coordination of the lower extremity. The orienteerers are asked to perform the exercises four times a week throughout the entire study period. The exercises are heel rises, runners pose, single leg stance and one-leg jumps with three difficult levels aiming to mainly improve lower extremity strength and neuromuscular function (online supplement). Each second week the exercises' difficulty level is increased.
  Interventions: Other: Exercise program
- Control (No Intervention): Normal training, no intervention

INTERVENTIONS:
Other: Exercise program — The orienteerers are asked to perform specific exercises four times a week throughout the entire study period. The exercises are heel rises, runners pose, single leg stance and one-leg jumps with three difficult levels aiming to mainly improve lower extremity strength and neuromuscular function. Each second week the exercises' difficulty level is increased.
  Arms: Intervention

SUMMARY:
The aim of this study is to investigate the effect a specific exercise program on the incidence of injuries in the lower extremity. 72 elite orienteerers, aged 18-40 years, are allocated to an intervention or control group. The intervention group performs four specific exercises, four times a week (10 minutes per session) in conjunction with normal training. Injury data are collected every second week using valid injury questionnaire distributed by text messages over 14 weeks. Primary outcome is number of substantial injuries in the lower extremity. Secondary outcomes are incidence of ankle sprains and the average substantial injury prevalence across the 10 weeks.

DETAILED DESCRIPTION:
The high physical load associated with running through uneven terrain contributes to that orienteerers are exposed to high injury risk, where the majority of injuries located in the lower extremities. Specific training programmes have been effective at reducing injury risk in sports. Yet, not trial has been conducted in elite orienteering. The aim of this study is to investigate the effect a specific exercise program on the incidence of injuries in the lower extremity. 72 elite orienteerers, aged 18-40 years, are allocated to an intervention or control group. The intervention group performs four specific exercises, with three difficult levels intensified every second week over the first four weeks, targeting strength, flexibility and coordination of the lower extremity. The exercises are completed four times a week (10 minutes per session) in conjunction with normal training. Injury data are collected every second week using valid injury questionnaire distributed by text messages over 14 weeks. Primary outcome is number of substantial injuries in the lower extremity. Secondary outcomes are incidence of ankle sprains and the average substantial injury prevalence across the 10 weeks. Participants will be recruited in January-February 2018. The intervention starts in February 2018 and data collection will be completed in June 2018. Data analyses are expected to be completed in October-November 2018.

Due to high injury risk and lack of injury prevention trials in orienteering, a RCT investigating the effect of a specific exercise program on the incidence of injuries in the lower extremity, is warranted. The results of this trial will be beneficial to orienteerers, clubs, federations and increase our understanding on how lower extremity injuries can be prevented in a physically challenging sport.

ELIGIBILITY:
Inclusion Criteria:

Adult elite orienteerers Aged 18-40 years Participating in the highest national orienteering league (Swedish League) Participant inclusion criteria - Age group: Adult Participant inclusion criteria - Gender: Both

Exclusion Criteria:

Injured adult elite orienteerers not able to perform baseline tests

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Lower extremity injury | March-June 2018 (10 weeks)
  Number of substantial injuries in the lower extremity

SECONDARY OUTCOMES:
Ankle sprain | March-June 2018 (10 weeks)
  Incidence of ankle sprains injuries
Substantial injury | March-June 2018 (10 weeks)
  The average substantial injury prevalence

CONTACTS AND LOCATIONS:
Overall Officials: Philip von Rosen, Study Chair — Karolinska Insitute
Locations (1):
- Karolinska Institutet, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Rosen P, Halvarsson B. Preventing lower extremity injury in elite orienteerers: study protocol for a randomised controlled trial. BMJ Open Sport Exerc Med. 2018 Apr 20;4(1):e000347. doi: 10.1136/bmjsem-2018-000347. eCollection 2018. PMID 29707231